CLINICAL TRIAL: NCT01963052
Title: A Phase 1 Study of the Safety and Pharmacokinetics of Escalating Doses of AGS15E Given as Monotherapy in Subjects With Metastatic Urothelial Cancer
Brief Title: ASG-15ME is a Study of Escalating Doses of AGS15E Given as Monotherapy in Subjects With Metastatic Urothelial Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGS15E-13-1
Record Dates: First submitted 2013-10-07; First posted 2013-10-16 (Estimated); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Urothelial Cancer
Keywords: Metastatic Urothelial Cancer; AGS15E; AGS15E-13-1; ASG-15ME; Pharmacokinetics of AGS15E
MeSH Terms: interventions — sirtratumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: AGS-15E Dose Escalation (Dose Levels 1-6) (Experimental): Subjects will receive a single 30 minute intravenous (IV) infusion of AGS15E once weekly for 3 weeks of every 4 weeks (Days 1, 8, and 15). A cycle is 4 weeks. Additional subjects may be enrolled for expansion of these dose levels to further evaluate the safety and efficacy, as recommended by a data review team (DRT).
  Interventions: Drug: AGS15E
- Part B: AGS-15E Cisplatin Therapy -ineligible Expansion (Experimental): Urothelial subjects who have not received any prior lines of therapy an who are unfit for Cisplatin therapy (Cis-ineligible) will receive a single 30 minute intravenous (IV) infusion of AGS15E once weekly for 3 weeks of every 4 weeks (Days 1, 8, and 15). A cycle is 4 weeks. Subjects will initially be dosed one dose level below the preliminary recommended phase 2 dose (RP2D).
  Interventions: Drug: AGS15E
- Part C: AGS15E Immune Checkpoint Inhibitor Treated Expansion (Experimental): Subjects previously treated with immune checkpoint inhibitors (CPI) in the metastatic setting will receive a single 30 minute intravenous (IV) infusion of AGS15E once weekly for 3 weeks of every 4 weeks (Days 1, 8, and 15). A cycle is 4 weeks. Subjects will be dosed at the RP2D.
  Interventions: Drug: AGS15E
- Part A: AGS15E Dose Expansion (Experimental): Subjects will receive a single 30 minute intravenous (IV) infusion of AGS15E once weekly for 3 weeks of every 4 weeks (Days 1, 8, and 15). A cycle is 4 weeks.
  Interventions: Drug: AGS15E

INTERVENTIONS:
Drug: AGS15E — intravenous (IV) infusion

SUMMARY:
The objectives of this study are to assess the safety, pharmacokinetics, immunogenicity and anti-tumor activity of AGS15E in subjects with metastatic urothelial cancer who failed at least one prior chemotherapy regimen for metastatic disease.

DETAILED DESCRIPTION:
All subjects will receive a single intravenous infusion of AGS15E once weekly for 3 weeks of every 4 weeks. A cycle is 4 weeks. Subjects will continue treatment until disease progression, intolerability of AGS15E, investigator decision, or consent withdrawal.

In subjects who discontinue therapy without documented disease progression and who still consent to study procedures, every effort should be made to continue monitoring their disease status by radiographic imaging until progression is documented, or new anticancer therapy, or death. All subjects will continue to be followed for survival until withdrawal of consent or study closure.

If assessed as complete response (CR) or partial response (PR) per local review a confirmatory scan will be performed no less than 4 weeks from previous scan and preferably at week 5. Tumor imaging should also be performed whenever disease progression is suspected.

Images will be sent to a central third party imaging vendor for an independent assessment per RECIST version 1.1. Although the imaging studies will be reviewed by a central third party imaging vendor in a retrospective fashion, all clinical decisions will be based on the interpretation of the investigator at the site treating the subject.

Post-Treatment Follow-up Progression Free Survival:

Subjects who discontinued study treatment for reasons other than radiographic disease progression will continue for a maximum of up to 12 months following the last dose of study drug until radiologically confirmed progression, initiation of a new anticancer therapy, death, loss to follow-up or withdraw consent for further follow-up, whichever of these events occurs first. The purpose of the post-treatment follow-up is to ascertain the duration of progression-free survival for all subjects enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Transitional Cell Carcinoma of the Urothelium (TCCU) (i.e., cancer of the bladder, renal pelvis, ureter, or urethra). Subjects with Urothelial Carcinoma with squamous differentiation or mixed cell types are eligible.
* Part A: Subject must have failed at least one prior chemotherapy regimen for metastatic disease and/or is unfit for cisplatin-based chemotherapy.
* Part B: Subject must not have received any prior lines of chemotherapy in the metastatic setting (prior treatment with immunotherapy is allowed).
* Part C (CPI-Treated Expansion): Subject must have received prior treatment with a CPI in the metastatic setting
* Subjects must have measureable disease according to RECIST (version 1.1).
* Part A and C: Subject must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Part B: Subject must have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
* Life expectancy of ≥ 3 months
* Adequate hematologic function
* Parts A and C: Renal function, as follows: serum creatinine ≤ 2.0 mg/dL, or measured 24 hour creatinine clearance of ≥ 45 mL/min
* Part B: Renal function, as follows: creatinine clearance estimate ≥ 15 mL/min and <60 mL/min by Cockcroft Gault equation adjusted for body weight
* Adequate liver function

Exclusion Criteria:

* Preexisting sensory neuropathy Grade ≥ 2 or motor neuropathy Grade ≥ 2
* Uncontrolled central nervous system metastases
* Use of any investigational drug within 14 days prior to the first dose of study drug
* Any anticancer therapy, including: small molecules, immunotherapy, chemotherapy, monoclonal antibody therapy, radiotherapy or any other agents to treat cancer (anti-hormonal therapy given as adjuvant therapy for early-stage estrogen receptor (ER) positive breast cancer is not considered cancer therapy for the purpose of this protocol)
* Subjects with Immunotherapy related adverse events requiring high doses of steroids (≥ 40 mg/day of prednisone) are not eligible
* Any P-gp inducers/inhibitors or strong CYP3A inhibitors within 14 days prior to the first dose of study drug
* History of thromboembolic events and/or bleeding disorders ≤ 14 days (e.g., deep vein thrombosis (DVT) or pulmonary embolism (PE)) prior to the first dose of study drug
* Active angina or Class III or IV Congestive Heart Failure (CHF) (New York Heart Association CHF Functional Classification System) or clinically significant cardiac disease within 12 months of study enrollment, including myocardial infarction, unstable angina, grade 2 or greater peripheral vascular disease, congestive heart failure, uncontrolled hypertension, or arrhythmias not controlled by outpatient medication
* Known HIV or AIDS
* Positive Hepatitis B surface antigen test
* Positive Hepatitis C antibody test
* Decompensated liver disease as evidenced by clinically significant ascites refractory to diuretic therapy, hepatic encephalopathy, or coagulopathy
* Known sensitivity to any of the ingredients of the investigational product AGS15E
* Major surgery within 28 days prior to first dose of study drug
* History of a primary invasive malignancy not listed in the inclusion criteria, which has not been in remission for at least 3 years. The following are exempt from the 3 year limit:

  * Non-melanoma skin cancer;
  * adenocarcinoma of the prostate that has been surgically treated with a post-treatment PSA that is undetectable;
  * cervical carcinoma in situ on biopsy or squamous intraepithelial lesion on Pap smear; and
  * definitively treated, stage I/II ER+ breast cancer
* Active infection requiring treatment ≤ 7 days before first dose of study drug
* History of uncontrolled diabetes mellitus or diabetic neuropathy
* Condition or situation which may put the subject at significant risk, may confound the study results, or may interfere significantly with subject's participation in the study
* Has ocular conditions such as:

  * Active infection or corneal ulcer (e.g., keratitis)
  * Monocularity
  * History of corneal transplantation
  * Contact lens dependent (if using contact lens, must be able to switch to glasses during the entire study duration)
  * Uncontrolled glaucoma (topical medications allowed)
  * Uncontrolled or evolving retinopathy, wet macular degeneration, uveitis, papilledema, or optic disc disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2013-11-14 (Actual); Primary Completion 2019-07-08 (Actual); Study Completion 2019-07-08 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | up to 36 months
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE): Concentration at the end of infusion (CEOI) | Days 1-4, 8, 15-18 and 22 of Cycle 1 and Days 1, 8, 15, 22 of Cycles 2 and 3, and Day 1 of subsequent cycles up to an average of 6 months
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE): Maximum observed concentration (Cmax) | Days 1-4, 8, 15-18 and 22 of Cycle 1 and Days 1, 8, 15, 22 of Cycles 2 and 3, and Day 1 of subsequent cycles up to an average of 6 months
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE): Trough concentration (Ctrough) | Days 1-4, 8, 15-18 and 22 of Cycle 1 and Days 1, 8, 15, 22 of Cycles 2 and 3, and Day 1 of subsequent cycles up to an average of 6 months
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE): Time to maximum concentration (Tmax) | Days 1-4, 8, 15-18 and 22 of Cycle 1 and Days 1, 8, 15, 22 of Cycles 2 and 3, and Day 1 of subsequent cycles up to an average of 6 months
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE): Partial area under the serum concentration-time curve after first dose and as appropriate (AUC0-7) | Days 1-4, 8, 15-18 and 22 of Cycle 1 and Days 1, 8, 15, 22 of Cycles 2 and 3, and Day 1 of subsequent cycles up to an average of 6 months
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE): Terminal or apparent terminal half-life (t1/2) | Days 1-4, 8, 15-18 and 22 of Cycle 1 and Days 1, 8, 15, 22 of Cycles 2 and 3, and Day 1 of subsequent cycles up to an average of 6 months
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE): Systemic clearance (CL) | Days 1-4, 8, 15-18 and 22 of Cycle 1 and Days 1, 8, 15, 22 of Cycles 2 and 3, and Day 1 of subsequent cycles up to an average of 6 months
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE): Volume of distribution at steady state (Vss) | Days 1-4, 8, 15-18 and 22 of Cycle 1 and Days 1, 8, 15, 22 of Cycles 2 and 3, and Day 1 of subsequent cycles up to an average of 6 months

SECONDARY OUTCOMES:
Incidence of Anti-Drug Antibody (ADA) | Up to 26 months
Tumor response | Up to 26 months
  Incidence of tumor response defined as either a complete response (CR) or partial response (PR) per RECIST criteria (version 1.1) that should be confirmed ≥ 28 days later
Objective response rate | Up to 26 months
  Defined as the percentage of subjects who experience a best response of either CR or PR in that cohort. CR and PR should be confirmed ≥ 28 days later
Disease control rate | Up to 26 months
  Defined as the percentage of subjects who experience a best response of CR, PR or stable disease (SD)
Progression free survival | Up to 36 months
  Time from the date of first infusion to the earliest date of documented disease progression per radiological evidence or death from any cause
Duration of response | Up to 36 months
  Time from the date of the first response CR or PR to the earliest date of disease progression or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Associate Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (11):
- United States (8):
  - Site US00006, Birmingham, Alabama
  - Site US00002, New Haven, Connecticut
  - Site US00001, Detroit, Michigan
  - Site US00003, St Louis, Missouri
  - Site US00009, Buffalo, New York
  - Site US00011, Pittsburgh, Pennsylvania
  - Site US00010, Nashville, Tennessee
  - Site US00008, Seattle, Washington
- Canada (3):
  - Site CA00004, Vancouver, British Columbia
  - Site CA00007, Hamilton, Ontario
  - Site CA00005, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Petrylak DP, Eigl BJ, George S, Heath EI, Hotte SJ, Chism DD, Nabell LM, Picus J, Cheng SY, Appleman LJ, Sonpavde GP, Morgans AK, Pourhosseini P, Wu R, Standley L, Croitoru R, Yu EY. Phase I Dose-Escalation Study of the Safety and Pharmacokinetics of AGS15E Monotherapy in Patients with Metastatic Urothelial Carcinoma. Clin Cancer Res. 2024 Jan 5;30(1):63-73. doi: 10.1158/1078-0432.CCR-22-3627. PMID 37861407